CLINICAL TRIAL: NCT02179918
Title: A PHASE 1B STUDY OF THE 4-1BB AGONIST PF-05082566 IN COMBINATION WITH THE PD-1 INHIBITOR MK-3475 IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study Of 4-1BB Agonist PF-05082566 Plus PD-1 Inhibitor MK-3475 In Patients With Solid Tumors (B1641003/KEYNOTE-0036)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B1641003; KEYNOTE-0036
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: interventions — utomilumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05082566 +MK-3475 (Experimental): PF-05082566 +MK-3475
  Interventions: Drug: PF-05082566; Drug: MK-3475

INTERVENTIONS:
Drug: PF-05082566 — Starting dose of 0.45 mg/kg q3wks IV, dose escalation
Drug: MK-3475 — 2 mg/kg q3wks, IV
  Other Names: pembrolizumab

SUMMARY:
This is a safety, pharmacokinetic and pharmacodynamic study designed to estimate the maximum tolerated dose (MTD), and determine the Recommended Phase 2 Dose (RP2D) of PF-05082566, a 4-1BB agonist monoclonal antibody (mAb), in combination with MK-3475, a PD-1 inhibitor in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced/metastatic solid tumor malignancy which has progressed on standard therapy or for which no standard therapy is available.
* Measurable disease per RECIST v1.1.
* Adequate bone marrow, renal and liver functioning

Exclusion Criteria:

* CNS primary malignancies, active seizure disorder or spinal cord compression, or carcinomatous meningitis.
* History of any of the following toxicities associated with a prior immunotherapy:

  * Grade 3 immune mediated adverse event that was considered related to previous immunotherapy and required immune suppressive therapy;
  * Grade 2 hepatic function related adverse event that persisted more than 1 week, was considered related to immunotherapy, or required treatment discontinuation or immunosuppressive therapy
* Any of the following within the 12 months prior to registration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
* History of or known presence of extensive, disseminated/bilateral or Grade 3 or 4 interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, or pulmonary fibrosis, but not including a history of prior radiation pneumonitis. Patients with clinically significant lung disease requiring oxygen therapy (eg, COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Research Administration Office, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - UCLA Oncology Center, Los Angeles, California
  - Smilow Cancer Center at Yale-New Haven Hospital, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1641003&StudyName=A%20Study%20Of%204-1BB%20Agonist%20PF-05082566%20Plus%20PD-1%20Inhibitor%20MK-3475%20In%20Patients%20With%20Solid%20Tumors%20%28B1641003/KEYNOTE-0036%29

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion at a dose of 0.45 mg/kg every 3 weeks (q3wks) on Day 1 of each dosing cycle. MK-3475 as a 30-minute intravenous infusion at a dose of 2 mg/kg q3wks started 30 minutes after completion of PF-05082566 infusion.
- PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion at a dose of 0.9 mg/kg q3wks on Day 1 of each dosing cycle. MK-3475 as a 30-minute intravenous infusion at a dose of 2 mg/kg q3wks started 30 minutes after completion of PF- 05082566 infusion.
- PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion at a dose of 1.8 mg/kg q3wks on Day 1 of each dosing cycle. MK-3475 as a 30-minute intravenous infusion at a dose of 2 mg/kg q3wks started 30 minutes after completion of PF- 05082566 infusion.
- PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion at a dose of 3.6 mg/kg q3wks on Day 1 of each dosing cycle. MK-3475 as a 30-minute intravenous infusion at a dose of 2 mg/kg q3wks started 30 minutes after completion of PF-05082566 infusion.
- PF-05082566 5 mg/kg + MK-3475 2 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion at a dose of 5 mg/kg q3wks on Day 1 of each dosing cycle. MK-3475 as a 30-minute intravenous infusion at a dose of 2 mg/kg q3wks started 30 minutes after completion of PF- 05082566 infusion.
Period: Overall Study
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Started | 5 | 3 | 3 | 3 | 9
Completed | 1 | 0 | 1 | 0 | 1
Not Completed | 4 | 3 | 2 | 3 | 8
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 4 | 1 | 1 | 2 | 6
Not completed — Other | 0 | 1 | 0 | 0 | 1
Not completed — Subject refused further follow-up | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were assigned to study treatment.
Groups:
- PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion at a dose of 0.45 mg/kg q3wks on Day 1 of each dosing cycle. MK-3475 as a 30-minute intravenous infusion at a dose of 2 mg/kg q3wks started 30 minutes after completion of PF-05082566 infusion.
- Total: Total of all reporting groups
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (15.4) | 62.0 (11.4) | 51.7 (22) | 54.7 (21) | 58.8 (19.4) | 58.0 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 2 | 4 | 9
  Male | 4 | 3 | 1 | 1 | 5 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 4 | 3 | 0 | 3 | 5 | 15
  Black | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 0 | 1 | 3
  Other | 0 | 0 | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT) of PF-05082566 in Combination With MK-3475
Description: Severity of adverse events (AEs) was graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs occurring during the DLT observation period that were attributable to one or both study drugs were classified as DLTs. 1) Hematologic: Grade 4 neutropenia; Febrile neutropenia, defined as absolute neutrophil count (ANC) <1000/mm3 with a single temperature of >38.3C(101F) or a sustained temperature of 38C (100.4F) for more than 1 hour; Grade>=3 neutropenic infection; Grade>=3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia. 2) Non hematologic: Grade>=3 toxicities (non-laboratory); Grade>=3 nausea, vomiting or diarrhea despite maximal medical therapy; Grade 4 aspartate aminotransferase (AST) and alanine aminotransferase (ALT). 3) Other (non-AST/ALT) non-hematologic Grade>=3 laboratory value. 4) Inability to complete 2 infusions of MK-3475 and PF-05082566 during the DLT observation period.
Time Frame: First 2 cycles of treatment up to 24 months
Population: The DLT evaluable set was a subset of the safety analysis set and included all participants who were eligible, received both study treatments and who either experienced a DLT during the first 2 cycles of PF-05082566 or completed the 2 cycles' DLT observation period.
Measure: Number; unit: Participants
Groups:
- Total: Sum across the participants from all arms. PF-05082566 was administered as a 1 hour intravenous infusion at a dose of 0.45 mg/kg, 0.9 mg/kg, 1.8 mg/kg, 3.6 mg/kg, 5 mg/kg, respectively and then the MK-3475 as a 30 minute intravenous infusion at a dose of 2 mg/kg was co-administrated.
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) and Treatment Emergent Adverse Events (TEAEs) by Maximum CTCAE Grade (All Causalities)
Description: An AE was any untoward medical occurrence in a clinical investigation subject administered a product or medical device, regardless of its causal relationship with study treatment. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Any events occurring following start of treatment or increasing in severity were counted as treatment emergent. The severity was graded by National Cancer Institute (NCI) CTCAE v.4.03. Grade 1 was mild AE. Grade 2 was moderate AE. Grade 3 was severe AE. Grade 4 was life-threatening consequences and urgent intervention AE. Grade 5 was indicated death related to AE.
Time Frame: Baseline up to 90 days after the last dose of study drug, approximately 27 months
Population: The safety analysis set was used, which was defined as all participants who received at least 1 dose of study drug. Participants were classified according to the study treatment actually received.
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  SAE | 2 | 0 | 1 | 2 | 5 | 10
  AE | 5 | 3 | 3 | 3 | 9 | 23
  Grade 1 | 0 | 1 | 2 | 1 | 0 | 4
  Grade 2 | 2 | 1 | 0 | 0 | 2 | 5
  Grade 3 | 2 | 1 | 1 | 1 | 7 | 12
  Grade 4 | 0 | 0 | 0 | 1 | 0 | 1
  Grade 5 | 1 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Treatment Emergent Adverse Events (TEAEs) by Maximum CTCAE Grade (PF-05082566-related)
Description: An AE was any untoward medical occurrence in a clinical investigation subject administered a product or medical device, regardless of its causal relationship with study treatment. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Any events occurring following start of treatment or increasing in severity were counted as treatment emergent. The severity was graded by NCI CTCAE v.4.03. Grade 1 was mild AE. Grade 2 was moderate AE. Grade 3 was severe AE. Grade 4 was life-threatening consequences and urgent intervention AE. Grade 5 was indicated death related to AE.
Time Frame: Baseline up to 90 days after the last dose of study drug, approximately 27 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  SAE | 0 | 0 | 0 | 0 | 0 | 0
  AE | 4 | 3 | 3 | 2 | 6 | 18
  Grade 1 | 1 | 3 | 2 | 1 | 1 | 8
  Grade 2 | 3 | 0 | 1 | 0 | 4 | 8
  Grade 3 | 0 | 0 | 0 | 1 | 1 | 2
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Treatment Emergent Adverse Events (TEAEs) by Maximum CTCAE Grade (MK-3475-related)
Description: as for outcome 3
Time Frame: Baseline up to 90 days after the last dose of study drug, approximately 27 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  SAE | 1 | 0 | 0 | 0 | 0 | 18
  AE | 4 | 3 | 3 | 2 | 6 | 1
  Grade1 | 1 | 3 | 2 | 1 | 1 | 8
  Grade 2 | 3 | 0 | 1 | 0 | 4 | 8
  Grade 3 | 0 | 0 | 0 | 1 | 1 | 2
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Treatment Emergent Adverse Events (TEAEs) by Maximum CTCAE Grade (Both-related)
Description: as for outcome 3
Time Frame: Baseline up to 90 days after the last dose of study drug, approximately 27 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  SAE | 0 | 0 | 0 | 0 | 0 | 0
  AE | 4 | 3 | 3 | 2 | 6 | 18
  Grade 1 | 1 | 3 | 2 | 1 | 1 | 8
  Grade 2 | 3 | 0 | 1 | 0 | 4 | 8
  Grade 3 | 0 | 0 | 0 | 1 | 1 | 2
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Test Values Meeting Categorical Summarization Criteria by Maximum CTCAE Grade (Hematology)
Description: The hematology laboratory test included: absolute neutrophil count, hemoglobin, platelet count, white blood cell with differential, coagulation panel, urinalysis and pregnancy test. Laboratory results were categorical summarized according to the NCI-CTCAE criteria version 4.03. The total number of participants with hematology laboratory test was assessed.
Time Frame: Baseline up to 28 days after the last dose of study drug, approximately 25 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  Anemia Grade 0-1 | 3 | 2 | 2 | 1 | 6 | 14
  Anemia Grade 2 | 2 | 1 | 0 | 1 | 2 | 6
  Anemia Grade 3-4 | 0 | 0 | 1 | 1 | 1 | 3
  Hemoglobin Increased Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Hemoglobin Increased Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Lymphocyte Count Increased Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphopenia Grade 0-1 | 1 | 2 | 1 | 1 | 2 | 7
  Lymphopenia Grade 2 | 2 | 0 | 2 | 0 | 5 | 9
  Lymphopenia Grade 3-4 | 2 | 1 | 0 | 2 | 2 | 7
  Neutrophils (Absolute) Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Neutrophils (Absolute) Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (Absolute) Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Grade 0-1 | 5 | 3 | 3 | 3 | 8 | 22
  Platelets Grade 2 | 0 | 0 | 0 | 0 | 1 | 1
  Platelets Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cells Grade 0-1 | 4 | 3 | 2 | 3 | 7 | 19
  White Blood Cells Grade 2 | 1 | 0 | 1 | 0 | 2 | 4
  White Blood Cells Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Laboratory Test Values Meeting Categorical Summarization Criteria by Maximum CTCAE Grade (Chemistries)
Description: The chemical laboratory test included: sodium, potassium, total calcium, creatinine, albumin, alanine aminotransferase, alanine aminotransferase, glucose, phosphorus, magnesium, total bilirubin, blood urea nitrogen, alkaline phosphatase, lactate dehydrogenase, immunoglobulin G, total protein, uric acid, thyroid function assessments, hepatitis B and C tests. Laboratory results were categorical summarized according to the NCI-CTCAE criteria version 4.03. The total number of participants with chemistry laboratory test was assessed.
Time Frame: Baseline up to 28 days after the last dose of study drug, approximately 25 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  Alanine Aminotransferase (ALT) Grade 0-1 | 5 | 3 | 3 | 3 | 8 | 22
  ALT Grade 2 | 0 | 0 | 0 | 0 | 1 | 1
  ALT Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase Grade 0-1 | 4 | 3 | 3 | 1 | 9 | 20
  Alkaline Phosphatase Grade 2 | 1 | 0 | 0 | 1 | 0 | 2
  Alkaline Phosphatase Grade 3-4 | 0 | 0 | 0 | 1 | 0 | 1
  Aspartate Aminotransferase (AST) Grade 0-1 | 4 | 3 | 3 | 3 | 8 | 21
  AST Grade 2 | 1 | 0 | 0 | 0 | 1 | 2
  AST Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (Total) Grade 0-1 | 5 | 2 | 3 | 3 | 8 | 21
  Bilirubin (Total) Grade 2 | 0 | 1 | 0 | 0 | 0 | 1
  Bilirubin (Total) Grade 3-4 | 0 | 0 | 0 | 0 | 1 | 1
  Creatinine Grade 0-1 | 4 | 2 | 3 | 2 | 7 | 18
  Creatinine Grade 2 | 1 | 1 | 0 | 1 | 2 | 5
  Creatinine Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Hypercalcemia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia Grade 0-1 | 3 | 2 | 3 | 1 | 8 | 17
  Hyperglycemia Grade 2 | 1 | 0 | 0 | 2 | 1 | 4
  Hyperglycemia Grade 3-4 | 1 | 1 | 0 | 0 | 0 | 2
  Hyperkalemia Grade 0 | 4 | 3 | 3 | 3 | 9 | 22
  Hyperkalemia Grade 2 | 1 | 0 | 0 | 0 | 0 | 1
  Hyperkalemia Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Hypermagnesemia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Hypernatremia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia Grade 0-1 | 3 | 3 | 1 | 1 | 8 | 16
  Hypoalbuminemia Grade 2 | 1 | 0 | 1 | 1 | 1 | 4
  Hypoalbuminemia Grade 3-4 | 1 | 0 | 1 | 1 | 0 | 3
  Hypocalcemia Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Hypocalcemia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia Grade 0-1 | 5 | 3 | 3 | 3 | 8 | 22
  Hypoglycemia Grade 2 | 0 | 0 | 0 | 0 | 1 | 1
  Hypoglycemia Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia Grade 0-1 | 5 | 3 | 3 | 2 | 8 | 21
  Hypokalemia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia Grade 3-4 | 0 | 0 | 0 | 1 | 1 | 2
  Hypomagnesemia Grade 0-1 | 5 | 3 | 3 | 3 | 9 | 23
  Hypomagnesemia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia Grade 3-4 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia Grade 0-1 | 4 | 3 | 2 | 2 | 8 | 19
  Hyponatremia Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia Grade 3-4 | 1 | 0 | 1 | 1 | 1 | 4
  Hypophosphatemia Grade 0-1 | 4 | 3 | 2 | 0 | 6 | 15
  Hypophosphatemia Grade 2 | 1 | 0 | 1 | 1 | 3 | 6
  Hypophosphatemia Grade 3-4 | 0 | 0 | 0 | 2 | 0 | 2

8. Secondary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Criteria of Potential Clinical Concern
Description: Vital sign summaries included all vital sign assessments from the on-treatment period. All vital sign parameters including blood pressure (BP) and weight were summarized using actual values and changes from baseline for each visit over time. The changes computed were the differences from baseline. The participants meeting criteria of potential clinical concern were judged by investigator.
Time Frame: Baseline up to 28 days after the last dose of study drug, approximately 25 months
Population: The safety analysis set included all participants who received at least 1 dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than 1 study treatment, the participant was classified according to the first treatment received.
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Shift From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status to Worst on Study
Description: The ECOG shift from baseline to highest score during the on-treatment period was summarized by treatment group.ECOG Performance Status included 0, 1, 2, 3, and 4 grades. Grade 1 was Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature. Grade 2 was Ambulatory and capable of all self care but unable to carry out any work activities.Up and about more than 50% of waking hours. Grade 3 was capable of only limited self care, confined to bed or chair more than 50% of waking hours. Grade 4 was completely disabled. Cannot carry on any self care. Totally confined to bed or chair.
Time Frame: Baseline up to 28 days after the last dose of study drug, approximately 25 months
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  ECOG Performance Status worst to 1 | 0 | 2 | 0 | 1 | 4 | 7
  ECOG Performance Status worst to 2 | 2 | 0 | 0 | 0 | 0 | 2
  ECOG Performance Status worst to 3 | 1 | 0 | 0 | 1 | 2 | 4
  ECOG Performance Status worst to 4 and 5 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-05082566
Description: Maximum PF-05082566 observed serum concentration.
Time Frame: During Cycle 5 on Day 1 at pre-dose, end of infusion, and at 2, 6, and 24 hours after the start of infusion, day 8 (168 hours) and day 15 (336 hours) after start of infusion
Population: The PK concentration analysis set was a subset of the safety analysis set and included participants who had at least 1 post-dose concentration measurement above the lower limit of quantitation (LLOQ) for PF-05082566 or MK-3475.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 4 | 1 | 3 | 3 | 4
µg/mL | 7.628 (25) | 18.70 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 29.80 (16) | 60.35 (39) | 95.57 (16)

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MK-3475
Description: Maximum MK-3475 observed serum concentration.
Time Frame: During Cycle 5 Day 1 at pre-dose; and end of infusion.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 4 | 1 | 3 | 2 | 3
ng/mL | 63350 (22) | 71300 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 61090 (7) | 51920 (NA) — Only 2 participants were analyzed, therefore the geometric coefficient of variation was not applicable. Individual subject values are 46000 and 58600 ng/mL, respectively | 62030 (32)

12. Secondary Outcome: Time for Cmax (Tmax) of PF-05082566
Description: Time to reach PF-05082566 maximum observed serum concentration.
Time Frame: as for outcome 10
Population: The PK parameter analysis set was a subset of the safety analysis set and included participants who had at least 1 of the PK parameters of interest for PF-05082566 or MK-3475.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 4 | 1 | 3 | 3 | 4
hour | 1.44 [1.00 to 1.98] | 5.40 [5.40 to 5.40] | 1.07 [1.03 to 2.03] | 1.08 [1.07 to 1.25] | 1.15 [1.00 to 6.00]

13. Secondary Outcome: Pre-dose Concentration During Multiple Dosing (Ctrough) of PF-05082566
Description: PF-05082566 pre-dose concentration during multiple dosing
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 4
µg/mL | 0.7489 (33) | 1.210 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 1.664 (35) | 5.167 (NA) — Only 2 participants were analyzed, therefore the geometric coefficient of variation was not applicable.Individual subject values are 4.32 and 6.18 µg/mL, respectively. | 7.796 (9)

14. Secondary Outcome: Pre-dose Concentration During Multiple Dosing (Ctrough) of MK-3475
Description: MK-3475 pre-dose concentration during multiple dosing
Time Frame: During Cycle 5 Day 1 at pre-dose; and end of infusion.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 4 | 1 | 3 | 3 | 4
ng/mL | 18460 (33) | 19200 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 20390 (15) | 11250 (78) | 17280 (46)

15. Secondary Outcome: Terminal Half-life （t½）of PF-05082566
Description: PF-05082566 terminal half-life
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 4
hour | 179.3 (24.338) | 173.0 (NA) — Only 1 participant was analyzed, therefore the standard deviation was not applicable. | 144.7 (31.628) | 174.5 (NA) — Only 2 participant were analyzed, therefore the standard deviation was not applicable. Individual subject values are 141and 208 hour, respectively. | 164.8 (49.564)

16. Secondary Outcome: Clearance (CL) of Study Drug of PF-05082566
Description: Clearance of PF-05082566
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 4
mL/hr/kg | 0.4120 (32) | 0.5000 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 0.5182 (41) | 0.3894 (NA) — Only 2 participants were analyzed, therefore the geometric coefficient of variation was not applicable.Individual subject values are 0.254 and 0.597 mL/hr/kg, respectively. | 0.4763 (25)

17. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-05082566
Description: PF-05082566 volume of distribution at steady state
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 4
mL/kg | 101.4 (45) | 112.0 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 104.0 (18) | 93.19 (NA) — Only 2 participants were analyzed, therefore the geometric coefficient of variation was not applicable. Individual subject values are 52.0 and 167 mL/kg, respectively. | 104.6 (13)

18. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Time Tau, the Dosing Interval, Where Tau = 504 Hours (21 Days) [AUCtau] for PF-05082566
Description: PF-05082566 area under the serum concentration-time curve (AUC) from time 0 to time tau, the dosing interval, where tau = 504 hours (21 days) (AUCtau)
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 4
µg•hr/mL | 1093 (32) | 1800 (NA) — Only 1 participant was analyzed, therefore the geometric coefficient of variation was not applicable. | 3477 (41) | 9253 (NA) — Only 2 participants were analyzed, therefore the geometric coefficient of variation was not applicable. Individual subject values are 6030 and 14200 µg•hr/mL, respectively. | 10480 (25)

19. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of PF-05082566
Description: ADA blood samples were assayed for anti-PF-05082566 antibodies using a validated analytical method in compliance with Pfizer (anti-PF-05082566) standard operating procedures (SOPs). ADA data was listed and summarized for PF 05082566 by dose. Negative ADA: titer<6.23; Positive ADA: titer>=6.23.Treatment-induced ADA = ADA developed de novo (seroconversion) following biologic drug administration. Treatment-boosted ADA = pre-existing ADA that were boosted to a higher level following biologic drug administration.
Time Frame: Pre-dose (Day 1), Cycles 1, 3, 5, 7, and subsequently pre-dose (Day 1) every 2 cycles up to Cycle 12, and every 4 cycles thereafter
Population: The immunogenicity analysis set was a subset of the safety analysis set and included participants who have at least 1 ADA sample collected for either PF-05082566 or MK 3475.
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  Pre-dose ADA | 0 | 0 | 0 | 1 | 1 | 2
  ADA Anytime | 4 | 3 | 2 | 3 | 5 | 17
  Treatment-induced ADA | 4 | 3 | 2 | 2 | 4 | 15
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0 | 0
  Overall ADA Incidence | 4 | 3 | 2 | 2 | 4 | 15

20. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of MK-3475
Description: ADA blood samples were assayed for anti-MK-3475 antibodies using a validated analytical method in compliance with Merck (anti-MK-3475) SOPs.
Time Frame: Pre-dose in Cycles 1, 3, 5, 7 and subsequently pre dose every 2 cycles up to Cycle 12 and every 4 cycles thereafter and 28 days, and during follow-up (3 months and 6 months after the end of MK-3475 treatment).
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Objective Tumor Response
Description: Objective response (OR) was defined as complete response (CR) or partial response (PR) according to RECIST version 1.1 from the date of first dose of study treatment until documented disease progression.CR = at least 2 determinations of CR at least 4 weeks apart and before progression; PR = at least 2 determinations of PR or better at least 4 weeks apart and before progression (and not qualifying for a CR); Progression of disease (PD) = progression<=12 weeks after the date of first dose of study treatment (and not qualifying for CR, PR, SD or non-CR/non-PD); Stable disease (SD) (applicable only to participants with measurable disease at baseline) = at least 1 SD assessment (or better)>=6 weeks after the date of first dose of study treatment and before progression (and not qualifying for CR or PR). Both CR and PR were confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met.
Time Frame: Baseline, at Week 9, and then every 6 weeks up to 90 days after the last dose of study drug, approximately 27 months. For those patients who achieved a confirmed PR or CR, tumor assessments could be conducted as clinically indicated.
Population: The full analysis set (FAS) included all participants who received at least 1 dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than 1 treatment the participant was classified according to the first treatment received.
Measure: Number; unit: Participants
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Participants
  Complete response | 0 | 0 | 1 | 0 | 1 | 2
  Partial response | 2 | 0 | 0 | 1 | 1 | 4
  Stable disease | 2 | 2 | 1 | 2 | 3 | 10
  Objective progression | 1 | 1 | 1 | 0 | 4 | 7
  Objective response rate (CR+PR) | 2 | 0 | 1 | 1 | 2 | 6

ADVERSE EVENTS:
Time Frame: Baseline up to 90 days after the last dose of study drug, approximately 27 months
Arm/Group | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg | PF-05082566 5 mg/kg + MK-3475 2 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/3 | 0/3 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/3 | 1/3 | 2/3 | 5/9
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg (N=5) | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg (N=3) | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg (N=3) | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg (N=3) | PF-05082566 5 mg/kg + MK-3475 2 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05082566 0.45 mg/kg + MK-3475 2 mg/kg (N=5) | PF-05082566 0.9 mg/kg + MK-3475 2 mg/kg (N=3) | PF-05082566 1.8 mg/kg + MK-3475 2 mg/kg (N=3) | PF-05082566 3.6 mg/kg + MK-3475 2 mg/kg (N=3) | PF-05082566 5 mg/kg + MK-3475 2 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 3
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Presbyoesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 3
Administration site reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 3
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 3 | 0 | 3
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 1 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to strategic reasons before any expansion cohort patient was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-07-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02179918/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02179918/SAP_001.pdf